CLINICAL TRIAL: NCT05562518
Title: GRACE-trial: a Randomized Active-controlled Trial for vulvovaGinal atRophy in breAst Cancer Patients on Endocrine Therapy.
Acronym: GRACE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BC-09638
Record Dates: First submitted 2022-02-07; First posted 2022-09-30 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Vulvovaginal Atrophy; Breast Cancer
Keywords: breast cancer; vulvovaginal atrophy; endocrine therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Estrogens; Dehydroepiandrosterone; Probiotics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Estrogen (Active Comparator): locally administered estrogen (oestriol)
  Interventions: Drug: Estrogen
- Dehydroepiandrosterone (Active Comparator): locally administered dehydroepiandrosterone (DHEA)
  Interventions: Drug: dehydroepiandrosterone
- Estrogen + probiotics (Active Comparator): locally administered estrogen (oestriol) + probiotics
  Interventions: Drug: Estrogen + probiotics
- Moisturizer (Active Comparator): locally administered hyaluronic acid
  Interventions: Drug: Moisturizer

INTERVENTIONS:
Drug: Estrogen — 1 vaginal ovule daily for three consecutive weeks, followed by 1 vaginal ovule 2 times per week
  Arms: Estrogen
Drug: dehydroepiandrosterone — 1 vaginal ovule daily
  Arms: Dehydroepiandrosterone
Drug: Estrogen + probiotics — 1 vaginal ovule daily for 12 consecutive days, followed by 1 vaginal ovule 2 times per week
  Arms: Estrogen + probiotics
Drug: Moisturizer — 1 vaginal ovule daily for 14 consecutive days, followed by 1 vaginal ovule every three days
  Arms: Moisturizer

SUMMARY:
In this prospective active-controlled randomized trial the investigators will assess for the first time ever the different local treatments of vulvovaginal atrophy in breast cancer patients on endocrine therapy. These patients are currently inadequately treated based on ignorance of possible treatment modalities and stigmatization of vulvovaginal atrophy.

DETAILED DESCRIPTION:
In this prospective active-controlled randomized trial the investigators will assess for the first time ever the different local treatments of vulvovaginal atrophy in breast cancer patients on endocrine therapy. These patients are currently inadequately treated based on ignorance of possible treatment modalities and stigmatization of vulvovaginal atrophy.

While current knowledge on comparative data of the local treatments of vulvovaginal atrophy is based on retrospective data or one-to-one comparisons, we will prospectively evaluate all different local treatments based on patient-reported outcome measurements. This new data is mandatory for increasing the awareness of physicians of the treatment possibilities of vulvovaginal atrophy in breast cancer patients. Together with the use of different communication channels towards patients, this combination will substantially contribute to the increase of quality-of-life of breast cancer patients with vulvovaginal atrophy.

The primary objectives in this trial are two-fold. The first primary objective addresses the efficacy of the different implemented treatment strategies based on patient-reported outcome measurements (PROMs). These PROMs will be implemented prior to treatment and after initiation of the implemented treatments (estrogen, DHEA, probiotics or moisturizer). By implementing repeated PROM assessment, longitudinal evaluation of symptom alterations due to the treatment can be objectified.

The second primary objective is the safety evaluation of the implemented treatments. This evaluation will be achieved by measuring the sex hormone concentrations systemically with repeated longitudinal measurements.

In this study, the investigators will measure sex hormone concentrations through high-sensitive assessments based on LC-MS/MS. Considering the ALARA (as low a reasonably achievable) principle in radiation safety, we could extrapolate this ALARA principle to the safety of the local hormonal treatment of vulvovaginal atrophy in breast cancer patients, where potential differences in increase of sex hormone concentrations between the different treatment modalities could be objectified. Despite previous literature that could not show increased recurrence of breast cancer, this finding will play an import role in the decision-making of treatment of vulvovaginal atrophy in breast cancer patients. As mentioned earlier, a direct comparison of these sex hormone concentrations for the different treatment modalities is currently lacking.

As translational secondary objective, the investigators aim to investigate the microbial alterations when using local treatment for vulvovaginal atrophy. Identification of these alterations will contribute in understanding the pathophysiology of vulvovaginal atrophy and may unravel changes caused by the local treatment and may create opportunities in the future for additive treatment or new therapeutic strategies to ameliorate the quality-of-life of breast cancer patients with vulvovaginal atrophy.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer patient
* current endocrine therapy (AI or SERM)
* postmenopausal status, defined by:

  * 12 months amenorrhoea or
  * 6 months amenorrhoe and FSH level of >40 mIU/mL or

    *>6 weeks after bilateral oophorectomy or
  * induced postmenopause (ovarian function suppression using GnRH-analogue)
* presence of one or more symptoms of vulvovaginal atrophy (dyspareunia, dryness, irritation)

Exclusion Criteria:

* a history of vulvar or vaginal surgery (Inclusion is possible after hysterectomy. For these subjects no microbiome sampling will be performed. Microbiome analysis is not performed for these subjects.)
* current other vulvar or vaginal disease
* recent use of antibiotics/antifungals/corticosteroids (less than 1 month)
* current use of vaginal hormonal treatment or vaginal moisturizer: inclusion is possible after a washout period of 4 weeks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 160 (Estimated)
Dates: Start 2022-03-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in symptoms and quality of life after implementation of treatment in a time frame of 12 weeks using the EQ5D-questionnaire. | 12 weeks
  Efficacy of the implemented treatments will be assessed based on patient-reported outcome measurements (PROM) that describe symptoms and quality-of-life.
  The first primary outcome will be based on assessment using the EQ5D-questionnaire.
  This endpoint will be assessed at three time points: at start, after 6 weeks, and at the end (after 12 weeks). The change in these PROMs will be evaluated over the predefined timeframe of 12 weeks.
  The EQ5D-questionnaire includes a scale describing the general health of the participant at the predefined times, using a metric scale from 0 to 100 (0 being the worst health and 100 being the best health).
Change in symptoms and quality of life after implementation of treatment in a time frame of 12 weeks using the FACT-ES questionnaire. | 12 weeks
  Efficacy of the implemented treatments will be assessed based on patient-reported outcome measurements (PROM) that describe symptoms and quality-of-life.
  The second primary outcome will be based on assessment using the FACT-ES-questionnaire.
  This endpoint will be assessed at three time points: at start, after 6 weeks, and at the end (after 12 weeks). The change in these PROMs will be evaluated over the predefined timeframe of 12 weeks.
  The FACT-ES consists of question with answer possibilities from 0 to 4 (with the higher the score, the better the quality of life).
Change in sex steroid hormone concentrations in a time frame of 12 weeks. | 12 weeks
  The change in concentration of sex steroid hormone concentration as a surrogate for safety be be evaluated by measuring the sex hormone concentrations systemically with repeated longitudinal measurements. This endpoint will be assessed at three time points: at start, after 6 weeks, and at the end (after 12 weeks). The following sex steroid hormone concentrations will be assessed: estrone, estradiol, DHEA-S, DHEA, testosterone, and dihydrotestosterone.

SECONDARY OUTCOMES:
Identification of vaginal microbial alterations after implementation of treatment. | 12 weeks
  The vaginal microbiome will be determined at start and after 12 weeks. Bacterial DNA will be extracted and the microbiota will be identified using cpn60 sequencing. The change in microbial profiles between the two timepoints will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Hans Verstraelen, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No